CLINICAL TRIAL: NCT06248164
Title: Relationship of Lifestyle Habits and Health Characteristics of Parents and Children: An Epidemiological Study
Brief Title: Relationship of Lifestyle Habits and Health Characteristics of Parents and Children
Status: Recruiting | Type: Observational
Sponsor: Universidade Estadual Paulista Júlio de Mesquita Filho (Other)
Responsible Party: Principal Investigator, Bruna Thamyres Ciccotti Saraiva, PhD, Universidade Estadual Paulista Júlio de Mesquita Filho
Other Study IDs: 59261422.2.0000.5402
Record Dates: First submitted 2023-11-27; First posted 2024-02-08 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Adult Fathers and Mothers; Children and Adolescents, Boys and Girls
Keywords: Family atmosphere; Lifestyle; Public health

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Children and adolescents (sons and daughters): The study will consist of children and adolescents from six years of age.
  Interventions: Other: No intervention
- Parents (mothers and fathers): The study will consist of children and adolescents from six years of age and at least one of their biological parents to be evaluated.

INTERVENTIONS:
Other: No intervention — We will not carry out any type of intervention, just observe the behaviors and health parameters of parents and children.
  Groups: Children and adolescents (sons and daughters)

SUMMARY:
Lifestyle habits and health characteristics (e.g., excess weight) acquired in childhood and adolescence have a good chance of being carried into adulthood. In this sense, seeking to understand which factors can influence these habits and/or characteristics is of paramount importance. One of these factors that can influence the health of children and adolescents are the lifestyle habits and characteristics of these young people's parents. One of the lifestyle habits that appears to be related between parents and children is physical activity. However, most studies analyze the practice of physical activity between parents and children only considering the practice of total physical activity, that is, not considering the different domains of physical activity [ i) physical efforts carried out in the work environment, occupations in the case of adults and in the school environment in the case of children and adolescents; ii) physical activities carried out during leisure time; iii) physical activities carried out in the form of active commuting], in addition to there being little information considering the different intensities of physical activity (light, moderate, vigorous and very vigorous). Another gap to be addressed is the relationship between other health variables between parents and children, including unhealthy lifestyle habits, such as smoking, eating disorders and symptoms of anxiety and depression, as well as adverse health conditions, such as the presence of chronic diseases. and overweight, would be different considering the parents' practice of physical activity, for example; whether the possible relationship between excess weight between parents and children would be similar in children of physically active parents when compared to children of insufficiently active parents. Therefore, the objective of the present study will be to verify whether the different domains and intensities of physical activity are related between parents and children, as well as to verify whether other lifestyle habits and health characteristics are related between parents and children, considering the levels of activity. physical status of parents (physically active and insufficiently active).

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescent over 6 years old.

Exclusion Criteria:

-

Ages: 6 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The project will be carried out with children and adolescents from six years of age. The project will be publicized through social media, such as Facebook, WhatsApp, Instagram and also through television and radio. Participants who are interested in participating in the project and appear at the FCT-UNESP premises; parents must sign the informed consent form authorizing their children to participate in the study, as well as parents must also sign the consent form also agreeing to participate in the study (since this project will evaluate the health parameters of parents and children). Furthermore, children and adolescents must sign a consent form agreeing to participate in the study.
Sampling Method: Probability Sample
Enrollment: 176 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective measure of physical activity | Baseline
  The objective measurement of physical activity will be performed using the Actigraph GT3X accelerometer (ActiGraph, LLC, Pensacola, FL, USA). Evaluated will remain with the equipment for five full days (three weekdays and two weekend days).
Subjective measure of physical activity | Baseline
  Physical activity in different domains will be assessed using the questionnaire by Baecke et al. (1982). This instrument assesses the practice of physical activity through 16 questions in the last twelve months considering physical effort at work (for adults) and at school (for children and adolescents), the practice of sports activities or systematic exercises during leisure time and activities occupation in free time. In the field of work or school (in the case of children and adolescents), issues relating to physical efforts carried out at work are investigated, such as: time spent sitting, standing and walking in the work environment, carrying weights, whether the subject being assessed sweats a lot at work and how tired you feel after a day of work. In the leisure domain, leisure-time physical activity is considered, such as exercising at the gym or playing sports.

SECONDARY OUTCOMES:
Practice of physical activity in childhood and adolescence | Baseline
  To evaluate the practice of physical activity in childhood (ages 7 to 10 years) and adolescence (11-17 years) two questions will be asked: whether they practiced any type of sport in these stages of life under the supervision of a teacher, with two alternatives of answer: yes or no.
Sedentary behavior (subjective measure) | Baseline
  To assess sedentary behavior, participants (parents and children) will answer the Sedentary Behavior Questionnaire (SBQ). It includes the domains of sedentary behavior (watching TV, playing video games and computer, sitting listening to music, sitting talking on the phone, working on the computer or bureaucratic tasks {e.g. answering emails}, playing a musical instrument, doing construction work art or crafts, sitting in a car, bus, or train) during the week and on weekends.
Sedentary behavior (objective measure) | Baseline
  To assess CS with direct measurement, participants will use the Actigraph GT3X (ActiGraph, LLC, Pensacola, FL, USA). The accelerometer data will be filtered, digitized and adjusted to a frequency of 30Hz with an interval (epoch) of 60 seconds. The accelerometer will be analyzed by ActiLife 6 software (ActiGraph, LLC, Pensacola, FL, USA). Data will be considered complete if the participant wears the accelerometer for at least 10 hours per day for 4 days. It will be used to characterize sedentary behavior when measuring <100 counts/min (< 1.5 METs). The outcome of interest will be the time spent in sedentary activity, the number of minutes per day, which will be converted into hours for the analyses, according to the cutoff point of Matthews et al. (2008).
Blood pressure | Baseline
  Blood pressure will be assessed using an Omron automatic blood pressure measuring device (Model HEM-742, Japan).
Height | Baseline
  Height will be measured standing up, with a fixed stadiometer and with individuals barefoot, will be displayed in centimeters.
Body mass | Baseline
  Body mass was measured using a digital scale, on which the individuals were barefoot and wearing light clothing, expressed in kilograms.
Body mass index | Baseline
  Based on body mass and height measurements, the body mass index (BMI) will be calculated by dividing the participant's weight by their height squared, expressed in kilograms per meter squared.
Waist circumference | Baseline
  Abdominal obesity will be determined by waist circumference, using an inextensible metallic tape, will be displayed in centimeters.
Autonomic Cardiac Modulation | Baseline
  The heart rate variability will be collected by means of the POLAR V800
Bone Mineral Density | Baseline
  The dual-energy X-ray absorptiometry technique (DEXA, Lunar DPX-NT; General Electric Healthcare, Little Chalfont, Buckinghamshire, United Kingdom) will be used to measure lean body mass in kilograms (kg) and bone mineral density (BMD ) in grams per square centimeter (g/cm2) of arms, legs, trunk, pelvis, spine and entire body. The equipment's own software will be used (GE Medical System Lunar, version 4.7). The analysis procedures were reported in a previous study by Saraiva et al. (2021). The machine's accuracy in terms of coefficient of variation was tested in a pilot study with 30 volunteers not involved in this study and resulted in an error of less than 1%. Both parents and children will undergo this assessment.
Quality of life - Adults | Baseline
  To assess HRQoL, the Medical Outcomes Study SF-36-Item Short Form Health Survey (SF-36) instrument was used. The SF-36 is made up of 36 items that cover eight domains regarding HRQoL: functional capacity, physical limitations, body pain, general perception of health, vitality, social aspects, emotional limitations, mental health and current perception of health in comparison a year ago. This instrument presents a final score from 0 to 100, where 0 represents the worst score and 100 represents the best score in relation to HRQoL (WARE et al., 1992).
Quality of life - Children and adolescents | Baseline
  Will be assessed using the KIDSCREEN-52 questionnaire. This instrument was developed in European countries to assess the health-related quality of life of children and adolescents (RAVENS-SIEBERER, et al., 2001). T
Anxiety and depression | Baseline
  The Hospital Anxiety and Depression Scale (HADS) will be used, which contains 14 multiple-choice questions, seven of which assess symptoms of anxiety and seven of depression. Each item can be scored from 0 to 3 and the maximum score is 21, for both anxiety and depression (ZIGMOND & SNAITH, 1983). This scale is also validated for use with children and young people (WHITE et al., 1999).
Stress | Baseline
  This aspect will be assessed in the parents of adolescents participating in the study using the Brazilian version of the Perceived Stress Scale (COHEN et al., 1983), validated by Siqueira Reis et al. (2010) which consists of 14 items about the frequency of feelings and thoughts related to events and situations that occurred in the last month, with seven items being negative (1, 2, 3, 8, 11, 12 and 14) and seven items being positive (4, 5, 6, 7, 9, 10, and 13). Each item is answered on a five-point Likert frequency scale, with 0=never and 4=very often. The stress score is constructed by adding the values answered in each of the items, with positive items being on an inverse scale (0=very often and 4=never). The total score varies from 0 to 56 points and the higher the score, the higher the stress level.
Musculoskeletal symptoms | Baseline
  The presence of musculoskeletal symptoms will be assessed using a questionnaire developed by Kuorinka et al. (1987) and validated for its use in the Brazilian population (PINHEIRO et al., 2002). This instrument assesses some musculoskeletal symptoms such as the presence of pain, tingling or numbness in different parts of the body (neck, shoulder, upper back, elbows, wrists/hands, lower back, hip/thigh, knees and ankles/feet ). It is noteworthy that this instrument is also validated for use with children and adolescents (LEGAULT et al., 2014). The intensity of pain and how long the participant has felt pain will also be assessed on a scale of zero to ten.
Quality of sleep | Baseline
  Will be assessed using the Mini-sleep Questionnaire (ZOMER et al. 2005), validated for the Portuguese language (FALAVIGNA et al. 2011), which consists of 10 questions with seven possible answers. (never= 1, very rarely= 2, rarely= 3, sometimes= 4, often= 5, very often= 6 and always= 7) and provides a dimensionless score (higher score, worse sleep quality). The final score generated by the instrument can be classified as: good sleep (score between 10 and 24 points), slightly altered sleep (score between 25 and 27 points), moderately altered sleep (score between 28 and 30 points) and very altered sleep ( score above 30 points). Subjects who have a score equal to or greater than 28 points will be classified as having altered sleep.
Sleep latency | Baseline
  Sleep latency will be investigated using the Pittsburg questionnaire (BUYSSE et al., 1989).
Eating habits | Baseline
  Eating habits will be verified through the frequency of weekly consumption of different foods based on the work of Block et al. (2000). The consumption of foods such as vegetables, fruits, cereals, dairy products, fried foods, sodium and sugary drinks (soft drinks), as well as stimulant (energy) and caffeinated drinks will be analyzed.

OTHER OUTCOMES:
Smoking | Baseline
  Smoking will be assessed using the following question: Do you smoke, have you smoked, or have you never smoked? If you smoke, how many cigarettes do you usually smoke per day, considering the last month? If you have smoked, how long have you smoked and how long have you stopped smoking?" Exposure to tobacco among non-smokers and ex-smokers will be assessed by the following question: "Do you have close contact with any smokers? Yes or no?"
Alcoholism | Baseline
  Alcohol consumption will be assessed by the weekly frequency of alcohol intake and the number of doses consumed. Adults who reported drinking alcoholic beverages with a frequency equal to or greater than 1-2 days a week with an intake of 1-2 drinks per day will be considered to have high alcohol consumption (each dose will correspond to 250 ml for beer and 40 ml for soft drinks distilled).
Economic condition | Baseline
  In determining the economic condition of families, the "Brazilian Economic Classification Criteria" established in 2011 by the Brazilian Association of Business and Research (ABEP) will be used, according to a database from a survey carried out in 2009. by the Brazilian Institute of Public Opinion and Statistics (ABEP, 2009).
Coronavirus | Baseline
  As the coronavirus may exert or have exerted influences on some of the variables investigated in this study (for example: mental health, cardiac autonomic modulation), participants will be asked: Have you been diagnosed with Covid-19? If so, how did your clinical condition evolve? Asymptomatic, mild symptoms, moderate symptoms (I needed medication), severe symptoms (I needed hospitalization), very serious symptoms (I needed intensive therapy).

CONTACTS AND LOCATIONS:
Locations (1):
- Diego Giulliano Destro Christofaro, Presidente Prudente, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No